CLINICAL TRIAL: NCT01803295
Title: Evaluating the Effect of Pre-TURBT Intravesical Instillation of Mitomycin C (MMC) Mixed With TC-3 Gel in Patients With Non Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Pre-TURBT TC-3 Gel Intravesical Instillation in NMIBC
Acronym: OPTIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-4M-CS-0002-0
Record Dates: First submitted 2013-02-21; First posted 2013-03-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Carcinoma of Urinary Bladder, Superficial
Keywords: Non Muscle Invasive Bladder Cancer; Intravesical instillation; Mitomycin C; Hydrogel Reverse thermal gelation; Drug retention; Urinary Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Mitomycin
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Diseases; Urologic Diseases | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40 mg MMC gel (Experimental): Device: TC-3 gel mixed with Mitomycin C (MMC) Six weekly intravesical instillations of 60 cc of TC-3 gel mixed with 40 mg MMC will be instilled using catheter.
  Other Name: MMC Gel
  Interventions: Device: 40 mg MMC gel
- Standard of care MMC mixed with water (Active Comparator): 40 mg MMC mixed with 40cc water. Six weekly intravesical instillations of 40 mg of MMC mixed with 40 cc of water will be instilled using catheter
  Interventions: Other: Standard of care MMC mixed with water
- 80 mg MMC gel (Experimental): Device: TC-3 gel mixed with Mitomycin C (MMC) Six weekly intravesical instillations of 60 cc of TC-3 gel mixed with 80 mg MMC will be instilled using catheter.
  Other Name: MMC Gel
  Interventions: Device: 80 mg MMC gel

INTERVENTIONS:
Device: 40 mg MMC gel — A reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature)for drug retention in the urinary bladder.
  Other Names: MMC-Gel
  Arms: 40 mg MMC gel
Other: Standard of care MMC mixed with water — Standard of care 40mg MMC mixed with water
  Arms: Standard of care MMC mixed with water
Device: 80 mg MMC gel — A reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature)for drug retention in the urinary bladder
  Other Names: MMC-Gel
  Arms: 80 mg MMC gel

SUMMARY:
In the proposed study the investigators aim to evaluate the effect of the standard of care dose (40mg) of MMC mixed with TC-3 gel (with sustained release mechanism on the drug) on low risk recurrent NMIBC lesions and to compare our findings to instillation with the standard mode of instillation- 40mg MMC in water in order to examine our hypothesis that MMC mixed with TC-3 gel will have at least non-inferior and even superior results over the standard instillation mode

The investigators believe that this study is of importance of several aspects:

1. It evaluates a new mode of bladder instillation that may bypass the drawbacks of the current instillation mode.
2. If proved effective this mode of treatment might save the need of TURBT performance and serve as a new mode of tumor ablation.
3. Even if proved partially effective this mode of treatment will diminish tumors size or number thus enable a more limited TURBT procedure.
4. This mode of treatment will enable immediate medical attendance to the patient's tumor recurrence without the waiting period (resulting from queues in the medical centers) for TURBT, which might improve the patient's prognostic outcome.
5. If this experimental treatment will prove to have a better ablative effect, this could be translated to a better prophylactic effect of tumor recurrence.

DETAILED DESCRIPTION:
Non-muscle-Invasive Bladder cancer is mainly treated by tumor resection (Trans Urethral Resection - TUR), followed by series of intravesical instillations of prophylactic chemotherapeutic drugs as Mitomycin C (MMC) or BCG. This treatment approach is limited due to rapid dilution the chemotheraputic drug by the incoming urine and clearance by urination.

TheraCoat core technology is based on a reverse thermal biodegradable gel (TC-3) (low viscosity at 5°C gel appearance at body temperature)for drug retention in the urinary bladder.

Prior to instillation, the TC-3 hydrogel, in a liquid state, is mixed with MMC.TC-3 mixed with MMC is instilled to the bladder by a catheter. Following gel insertion to the bladder, the gel solidifies and forms a drug reservoir inside the bladder. Upon contact with urine the gel dissolves and is cleared out from the bladder.

Intravesical MMC instillation using TheraCoat gel is expected to increase treatment efficiency due to prolongation of treatment duration and consequently improving bladder exposure to MMC.

Treatment Protocol - Immediately following baseline cystoscopy and tumor diagnosis and patient undergoes 6 weekly instillations followed by 2-4 weeks healing period.

1st Follow-Up Visit (Pre-Scheduled TURBT Visit): The patient will undergo a second Cystoscopy to compare to the Baseline status and after that a follow-up period: 3,6,9,12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 21 years of age or older.
2. Patient has signed Informed Consent Form and is willing and able to abide by the protocol.
3. Naïve or recurrent low grade (LG) NMIBC tumor
4. Recurrent patients - Single or multiple tumors
5. Naive patients - 2 tumors or above
6. No prior history of HG and/or T1 in the past 5 years.
7. No prior history of Tis
8. At least one Tumor ≥ 1 mm as evaluated visually by the investigator.
9. Largest tumor diameter ≤ 30 mm as evaluated visually by the investigator
10. Cystoscopic appearance of papillary Low grade tumor
11. No active urinary tract infection as confirmed by urine culture
12. If the patient is a female of childbearing potential , she is using two acceptable & effective methods of contraception , until 6 months post treatment
13. If the patient is a male he should use a condom during intercourse, for at least 48 hours post each instillation
14. If the patient is a male that has a partner that is a female of childbearing potential, he should be advised to use two acceptable & effective methods of contraception until 6 months post treatment.

Exclusion Criteria:

1. Carcinoma In Situ (CIS).
2. "High Grade" urine cytology which is conclusive for HG.
3. "High Grade" tumor results in cold cup biopsy.
4. Tumor located in prostatic urethra.
5. Previous systemic chemotherapy in the last 2 years or pelvic radiotherapy.
6. Pregnant or breastfeeding patient.
7. Previous treatment with BCG within the last 12 months.
8. The patient did not have at least 3 months cystoscopically confirmed tumor-free interval between the last TURBT to current tumor recurrence.
9. Treatment with full course of intravesical chemotherapy within the 3 last months.
10. The patient has/had any bladder tumor with histology other than TCC.
11. Known contraindication or hypersensitivity to MMC or gel.
12. The patient has a known history of upper urinary tract urothelial carcinoma, or Renal Cell carcinoma or other renal cancer.
13. The patient has a known urinary retention which, according to the investigator's opinion, might lead to avoid patient receiving the treatment.
14. The patient has a bleeding disorder or a screening platelet count <50X109/L.
15. The patient has screening hemoglobin <10 mg/dL.
16. The patient has a condition or a concurrent severe and/or uncontrolled medical or psychiatric disease (e.g. uncontrolled diabetes, compensated congestive heart failure (NYHA III and over), myocardial infarction within 6 months of study, unstable or uncontrolled hypertension or an active uncontrolled infection), which could compromise participation, compliance with scheduled visits and/or completion.
17. The patient participated in an investigational interventional study within the past 90 days.
18. The patient has documented sever vesico-ureteral reflux or an indwelling ureteral stent.
19. The patient has the tumor in the bladder diverticulum.
20. The patient participated in a prior TheraCoat's trial with MMC and TC-3

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
ablative effect of pre-TURBT intravesical instillations of the treatments on The bladder lesion(s) of NMIBC patients | 2 years
  Cystoscopic and pathological effect (evaluated during TUR-BT visit) of pre-TURBT intravesical instillations with 40 mg of MMC mixed with 60cc TC-3 Hydrogel on bladder lesion(s) of NMIBC patients. At To, which is the time of identification of a recurrent tumor by cystoscopy, the number, size and location of the lesions will be documented and photographed. Each tumor size will be evaluated by photographing a ureter catheter adjacent to the tumor. Since the ureter catheter diameter is a pre-known variable, the tumor diameter can be calculated using specific software developed for study purposes. Photography of the tumor with a pre-known diameter ureter catheter will be performed during the same cystoscopy as described above and will be evaluated by a central clinic for uniformity of measurements, and the results of these measurements will serve for the post study evaluation of the change in tumor diameter
Number of Participants with Adverse Events as a Measure of Safety and Tolerability rate. | 2 years
  Demonstration of Pre-TURBT TC-3 gel-MMC instillation safety and adverse event rate.Adverse events will be defined as any adverse change in health or side effect that occurs in the clinical trial participant while the patient is receiving the treatment or until the completion of the post-treatment follow-up cystoscopy.

OTHER OUTCOMES:
Comparison of the cystoscopic and pathological effect between the 2 groups. | 2 years
  • Comparison of the cystoscopic and pathological effect of pre-TURBT instillations with MMC mixed with TC-3 Hydrogel on bladder lesion(s) to that of pre-TURBT MMC in water instillation groups
• Comparison of one year tumor recurrence rate between both treatment groups | 2 years
• Demonstration that blood levels of MMC following Pre-TURBT TC-3 gel-MMC instillation are below the toxic level (400ng/ml) known in the art for IV MMC administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fred Witjes, Prof, Principal Investigator — Radboud University Nijmegen Medical Centre, Department of Urology Geert Grooteplein South 10 (659), Nijmegen; Stenzl, Prof., Principal Investigator — Tübingen Universitätsklinik für Urologie
Locations (13):
- Israel (7):
  - Carmel Medical Center of Haifa, Department of Urology, Haifa
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center of Holon, Department of Urology, Holon
  - Meir medical center, Kfar Saba
  - Galil Maaravi Medical Center of Nahariya, Department of Urology, Nahariya
  - Rabin Medical Center of Petah Tikva, Department of Urology, Petach Tikvah
  - Ziv Medical Center, Safed
- Italy (3):
  - Vita Salute University, San Raffaele Hospital of Milan, Department of Urology, Milan
  - S. Andrea Hospital of Rome, Department of Urology, Rome
  - Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
- Spain (2):
  - Fundacio Puigvert, Barcelona
  - Hospital Universitario Infanta Sofìa of Madrid, Department of Urology, Madrid
- Hôpital HUG of Geneva, Department of Urology, Geneva, Switzerland